CLINICAL TRIAL: NCT01632202
Title: The Role of Seprafilm Bioresorbable Slurry in the Prevention of Intrauterine Synechiae in Patients Undergoing Hysteroscopic Myomectomy
Brief Title: Seprafilm Slurry in the Prevention of Uterine Scarring in Patients Undergoing Hysteroscopic Myomectomy
Acronym: Seprafilm
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: No subjects were recruited at the Weill Cornell site.
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AAAF2293
Record Dates: First submitted 2012-06-28; First posted 2012-07-02 (Estimated); Results first posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Intrauterine Adhesions
Keywords: submucosal myomas; intrauterine adhesions; hysteroscopic myomectomy; seprafilm
MeSH Terms: conditions — Gynatresia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Seprafilm Slurry (Active Comparator): The investigators hypothesize that by placing a slurry of Seprafilm in the intrauterine cavity and creating a temporary physical barrier between the walls of the uterus, that we will be able to prevent iatrogenic intrauterine adhesions. Given that approximately 24 to 48 hours after placement, the membrane becomes a hydrated gel that is slowly resorbed within one week, we anticipate that the patient will have minimal to no discomfort; since no physical device is being left in the endometrial cavity, the uterus will not be contracting more than it does in its normal postoperative state.
  Interventions: Device: Seprafilm
- Placebo (Placebo Comparator): For those randomized not to receive Seprafilm slurry, a syringe will be filled with 25ml of sterile saline.
  Interventions: Device: Sterile Saline Solution

INTERVENTIONS:
Device: Seprafilm — Seprafilm Adhesion Barrier (membrane) is a sterile, bioresorbable, translucent adhesion barrier composed of two anionic polysaccharides, sodium hyaluronate (HA) and carboxymethylcellulose (CMC). Together, these biopolymers have been chemically modified with the activating agent 1-(3-dimethylaminopropyl) -3- ethylcarbodiimide hydrochloride (EDC).
  Arms: Seprafilm Slurry
Device: Sterile Saline Solution — For those randomized not to receive Seprafilm slurry, a syringe will be filled with 25ml of sterile saline.
  Arms: Placebo

SUMMARY:
Seprafilm is an FDA-approved temporary bioresorbable barrier that physically separates opposing tissue surfaces. The physical presence of the membrane separates adhesiogenic tissue while the normal tissue repair process takes place. When used in the abdominopelvic cavity, it has been shown to reduce the incidence of adhesions.

The intrauterine cavity is a potential space where the walls of the uterus are collapsed upon itself in the normal state. It has been demonstrated that the trauma of removing a submucosal fibroid with electrocautery exposes the uterus to great potential for intrauterine adhesions since the raw charred surface is directly opposed to the opposite endometrial surface. Previous studies have shown that the placement of hyaluronic acid in the intrauterine cavity after a myomectomy is not only safe, but also decreases the incidence of intrauterine adhesions.

The investigators hypothesize that by placing a slurry of Seprafilm in the intrauterine cavity and creating a temporary physical barrier between the walls of the uterus, that they will be able to prevent iatrogenic intrauterine adhesions. Given that approximately 24 to 48 hours after placement, the membrane becomes a hydrated gel that is slowly resorbed within one week, the investigators anticipate that the patient will have minimal to no discomfort; since no physical device is being left in the endometrial cavity, the uterus will not be contracting more than it does in its normal postoperative state.

DETAILED DESCRIPTION:
The investigators will conduct a randomized controlled trial (RCT) involving patients at NewYork Presbyterian Hospital-Columbia University Medical Center and Weill Medical College of Cornell University. The investigators will enroll 328 pre- menopausal patients (>18years) with documented submucosal myomas undergoing hysteroscopic myomectomy with monopolar resection in this study.

The investigators anticipate that approximately 30% of the patients undergoing myomectomy will form intrauterine adhesions and that administration of the Seprafilm slurry will reduce the incidence to approximately 15%.

Patients will be queried on post-operative days 1, 7, and 30 for pain/discomfort and the degree of intrauterine adhesions will be assessed after the patient's second menses (75-90 days post procedure).

ELIGIBILITY:
Inclusion Criteria:

* Reproductive aged women: Age 18-48 years old
* Non-pregnant
* Otherwise healthy
* Regular menstrual cycle
* Documented submucosal myomas (one or more)
* Undergoing hysteroscopic myomectomy
* Patients must have signed an informed consent.

Exclusion Criteria:

* Age < 18 or in menopause
* Undergoing a second uterine surgical procedure
* Other significant uterine pathology (including but not limited to adhesions, septae, or cancerous lesions)
* Hysteroscopic evidence of synechiae at the time of the procedure
* Surgeries complicated by excessive bleeding; defined by estimated blood loss > 100cc given that the presence of excessive bleeding may predispose a patient to the formation of intrauterine adhesions
* Surgeries complicated by uterine perforation
* Surgeries complicated by postoperative intrauterine infection given that infection may predispose a patient to the formation of intrauterine adhesions (If these patients received Seprafilm Slurry, they will continue to be followed for safety monitoring)

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rogerio A Lobo, MD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Weill Medical College of Cornell University, New York, New York
  - Columbia University Medical Center, New York, New York

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 11 signed a consent form, but only 8 were randomized.
Period: Overall Study
Arm/Group | Seprafilm Slurry | Placebo
Started | 1 | 7
Completed | 1 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Seprafilm Slurry | Placebo | Total
Number analyzed (Participants) | 1 | 7 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 7 | 8
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 7 | 8
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 1 | 3 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Presence of Iatrogenic Intrauterine Adhesions
Description: Number of Subjects with iatrogenic intrauterine adhesions. Evidence of uterine scarring will be evaluated by a 3D sonohysterogram.
  A 3D sonohysterogram will be performed in the standard fashion in our ultrasound department by a blinded practitioner. The degree of adhesive disease will be scored by standard convention as:
  * Absent Adhesive Disease: no presence of intrauterine adhesions
  * Mild Adhesive Disease: cavities that are less than or equal to 30% affected
  * Moderate Adhesive Disease: cavities that are greater than 30% but less than or equal to 60% affected
  * Severe Adhesive Disease: cavities that are greater than 60% affected
Time Frame: 2- 3 months after surgery
Population: Only 5 out of the 8 enrolled completed the 3D sonohysterograms and therefore were the only ones included in the data analysis for the primary outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Seprafilm Slurry | Placebo
Number analyzed (Participants) | 1 | 4
Participants | 0 | 0

2. Secondary Outcome: Pregnancy Within 12 Months of Treatment
Description: Number of pregnancies within 12 months of treatment. In order to determine if Seprafilm helps improve pregnancy rates we will be conducting an additional follow-up phone call up to 12 months from the day of sonohysterogram. In women who have wished to get pregnant we will ask if they have been trying to get pregnant and if they have gotten pregnant. Participation in this follow up call is optional.
Time Frame: Up to 12 months after surgery
Population: Only 3 out of the 8 randomized completed the fertility follow up. There were 2 subjects (1 in the treatment arm and 1 in the placebo arm) who were not actively trying to get pregnant, and therefore did not complete the fertility follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Seprafilm Slurry | Placebo
Number analyzed (Participants) | 1 | 2
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Post-operative Day 1, Post-operative Day 7, and Post-operative Day 30
Arm/Group | Seprafilm Slurry | Placebo
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/7
Other Adverse Events (participants affected / at risk) | 1/1 | 7/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Seprafilm Slurry (N=1) | Placebo (N=7)
Fever (General disorders) | 1 | 1
Flu (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pelvic Pain (General disorders) | 0 | 3
Uterine Cramps (Reproductive system and breast disorders) | 1 | 5
Vaginal Bleeding (Reproductive system and breast disorders) | 0 | 6
Vaginal Discharge (Reproductive system and breast disorders) | 1 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes